CLINICAL TRIAL: NCT06865833
Title: Non-Medication Methods to Relieve Adolescents with Somatoform Disorders
Acronym: Tai Chi Ados
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP232535
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Somatoform Disorders in Adolescents
Keywords: Chronic somatoform disorders; Somatic symptoms; Adolescent medicine; Tai Chi for chronic pain; Psychosomatic disorders; Mental health in adolescents
MeSH Terms: conditions — Medically Unexplained Symptoms; Psychophysiologic Disorders | interventions — Tai Ji

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adolescents with Chronic Somatoform Disorders: This cohort consists of adolescents aged 12 to 19 years who are experiencing chronic somatoform disorders, which involve persistent physical symptoms (such as abdominal pain, headaches, and fatigue) without an identifiable medical cause. These symptoms often lead to frequent medical consultations, school absenteeism, and emotional distress such as anxiety and depression.
  The intervention of interest in this study is a series of Tai Chi and relaxation workshops. These workshops will be held once a week for 5 consecutive weeks, with each session lasting 1 hour and 15 minutes. The goal is to evaluate the impact of Tai Chi and relaxation on reducing somatoform symptoms, alleviating pain, improving mood, reducing anxiety and depression, and enhancing overall quality of life. The study will assess changes in these outcomes before and after the intervention, using various questionnaires and clinical assessments.
  Interventions: Other: Tai Chi and Relaxation Intervention

INTERVENTIONS:
Other: Tai Chi and Relaxation Intervention — This Tai Chi and Relaxation Intervention specifically targets adolescents with chronic somatoform disorders, utilizing a combination of mind-body practices designed to reduce pain and alleviate psychological distress. The intervention is distinct in the following ways:
  Target Population: It focuses specifically on adolescents aged 12-19 years experiencing unexplained physical symptoms, such as chronic pain, headaches, and fatigue, that are not attributable to any identifiable medical condition.
  Non-pharmacological Approach: Unlike traditional medical treatments that may involve medications or invasive procedures, this intervention is entirely non-medical, aiming to address both the physical and psychological aspects of chronic somatoform disorders without using drugs.
  Structured Workshops: The intervention consists of weekly Tai Chi and relaxation workshops (1 hour 15 minutes per session) over a 5-week period. The approach emphasizes gentle, controlled movements, relaxation techniqu

SUMMARY:
This research aims to investigate the effects of Tai Chi and relaxation techniques on adolescents (12-19 years old) with chronic somatoform disorders. These disorders are characterized by unexplained physical symptoms, such as abdominal pain and headaches, that cannot be linked to any identifiable medical condition. Adolescents with these disorders often experience frequent medical consultations, hospitalizations, and a negative impact on their daily lives, including school attendance, social interactions, and family relationships.

Tai Chi, a non-medicinal mind-body practice, has shown promise in reducing chronic pain, stress, and anxiety in both children and adults. Given its non-violent, accessible nature, Tai Chi is an appealing option for adolescents experiencing somatoform symptoms. It is believed that Tai Chi can help alleviate physical pain, manage stress, and improve mood, thus enhancing the adolescents' overall quality of life.

The main objective of this study is to quantify the changes in somatoform symptoms, pain levels, medication use, healthcare visits (including emergency consultations), school absenteeism, and the overall quality of life before and after five weeks of Tai Chi sessions. Secondary objectives include evaluating the reduction of anxiety and depression through standardized questionnaires, such as the HAD scale. Additionally, the study will gather qualitative data to assess the motivations, benefits, and barriers to practicing Tai Chi among the adolescents.

The research will involve adolescents from the Trousseau Hospital's adolescent medicine unit. Data will be collected prospectively, providing important insights that may pave the way for future randomized controlled trials. This study hopes to offer a new, non-medical approach to managing chronic somatoform disorders and improving the well-being of adolescents affected by them.

DETAILED DESCRIPTION:
This research is designed to evaluate the potential benefits of Tai Chi and relaxation techniques in alleviating symptoms of chronic somatoform disorders in adolescents aged 12-19 years. Somatoform disorders are characterized by the presence of physical symptoms-such as abdominal pain, headaches, or fatigue-that do not have an identifiable organic cause. These disorders are particularly common among adolescents, with at least 10% of this age group experiencing unexplained physical complaints. These symptoms often lead to frequent medical consultations, including emergency visits, hospitalizations, and significant disruptions to the adolescents' daily lives, including their school performance, social relationships, and family dynamics.

In addition to the functional impairments caused by these symptoms, chronic somatoform disorders can also be associated with anxiety and depression, which can exacerbate the physical complaints. While traditional medical treatments, including medication, are commonly used to manage these symptoms, many adolescents continue to experience persistent issues, revealing the limitations of conventional treatments. As a result, non-medication methods are being increasingly explored to address the psychological and physical aspects of these disorders.

Tai Chi, a traditional Chinese martial art that combines slow, deliberate movements with deep breathing and mental focus, has shown promise in reducing chronic pain, improving stress management, and enhancing mental well-being in various populations. In particular, Tai Chi has been used effectively in adults to manage chronic pain and stress, in children to reduce anxiety, and in students to improve overall physical and psychological well-being. Given its non-violent nature and focus on mind-body integration, Tai Chi could offer an engaging and accessible therapeutic option for adolescents.

The primary aim of this research is to assess the evolution of somatoform disorders in adolescents before and after a series of Tai Chi sessions. This will be done by evaluating changes in various factors, including somatoform symptoms, pain intensity, medication use, healthcare visits (emergency consultations and hospitalizations), school absenteeism, anxiety, depression, and overall quality of life. The study will provide quantitative data on the effectiveness of Tai Chi in addressing these issues, with the goal of preparing for a future randomized controlled trial to formally assess the intervention's effectiveness.

Main Objective:

To quantify the changes in somatoform symptoms in adolescents receiving Tai Chi intervention. This objective is primarily descriptive and aims to provide precise, standardized data on the evolution of symptoms before and after the intervention. This data will be essential for planning future trials.

Secondary Objectives:

Pain Assessment: Changes in pain levels will be measured using a self-reported numerical pain scale (0-10) and by assessing other clinical signs associated with somatoform symptoms.

Medication Consumption: Evaluation of changes in the amount and type of medication used by the adolescents for managing pain or related symptoms.

Healthcare Utilization: Changes in the number of consultations, emergency visits, and hospitalizations related to somatoform disorders will be tracked.

School Absenteeism: The number of school days missed due to somatoform symptoms will be assessed through self-reported questionnaires.

Anxiety and Depression: The Hospital Anxiety and Depression (HAD) scale will be used to assess changes in anxiety and depression levels before and after the intervention.

Quality of Life: The SF-36 questionnaire will be used to evaluate changes in the adolescents' quality of life, focusing on physical and emotional well-being.

Qualitative Assessment: A brief qualitative questionnaire will be administered to explore the adolescents' perceptions of Tai Chi, including motivations to participate, benefits, and any barriers to practice.

Study Design:

The research will involve adolescents from the adolescent medicine unit at Trousseau Hospital. Participants will be recruited during medical consultations, and their consent or parental consent will be obtained. The adolescents will participate in five weekly Tai Chi sessions, each lasting 1.5 hours. The sessions will be led by Dr. Luce Condamine, a pediatrician who is trained and certified in Tai Chi, ensuring that the practice follows the standard protocols for this therapeutic approach.

The Tai Chi sessions will be structured to integrate both the physical movements and relaxation techniques, aiming to reduce pain, improve mental health, and foster better body awareness among the participants. Each session will include a combination of gentle movements, deep breathing, and mindful relaxation.

Assessment Tools:

CSI-24 (Somatization Inventory): The primary evaluation tool will be the CSI-24, which is a self-report scale assessing the severity of somatic symptoms experienced over the previous two weeks.

Numerical Pain Scale (0-10): To assess pain intensity. Medication Use (DCI): Medication consumption will be tracked, including dosage and frequency.

Healthcare Visits: Number of medical consultations, emergency visits, and hospitalizations will be recorded.

School Absenteeism: Number of missed school days will be tracked through self-reports.

HAD Scale: This scale measures anxiety and depression, with scores ranging from 0 to 21, categorizing the severity of symptoms.

SF-36 Questionnaire: A standardized tool used to measure overall quality of life, including both physical and mental health components.

Qualitative Questionnaire: Questions about the adolescents' experiences with Tai Chi and any perceived benefits or challenges will be included.

Data Collection and Analysis:

Data will be collected before and after the intervention (after the five Tai Chi sessions). The study will provide a prospective evaluation of the changes in the adolescents' symptoms and well-being. These data will be analyzed to identify any significant differences in somatoform symptoms, pain levels, medication use, healthcare visits, school absenteeism, anxiety, depression, and quality of life.

Ethical Considerations:

The study will adhere to ethical guidelines, ensuring informed consent is obtained from all participants or their legal guardians. The intervention does not pose any physical or psychological risks, and participation is voluntary. The data collected will be kept confidential and used solely for research purposes.

Conclusion:

This study aims to explore Tai Chi as a potential non-medication intervention for managing chronic somatoform disorders in adolescents. The results will provide valuable insights into the effectiveness of Tai Chi in improving somatoform symptoms, reducing pain, enhancing mental health, and improving overall quality of life. If successful, this approach could offer an accessible, non-invasive treatment option for adolescents struggling with somatoform disorders.

ELIGIBILITY:
nclusion Criteria:

* Adolescents aged between 12 and 19 years
* Somatic or somatoform complaints
* Understanding of instructions as assessed by the investigator
* Physically able to practice Tai Chi
* Patients/parents informed and not opposed to the research

Exclusion Criteria:

* Inability to participate in a group as assessed by the investigator Refusal to participate Any difficulty in understanding or reading French that may prevent the execution of the protocol, as assessed by the investigator Patient deprived of liberty or under judicial protection (guardianship, curatorship, legal safeguard)

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents consulting at Trousseau Hospital (ages 12-19) in the adolescent medicine unit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-10-04 (Estimated); Study Completion 2025-10-04 (Estimated)

PRIMARY OUTCOMES:
CSI-24 Score (Somatization Inventory 24) | 5 weeks
  he CSI-24 is a self-reported scale that assesses the intensity of 24 somatic symptoms experienced by adolescents over the past two weeks. Higher scores indicate more severe somatic symptoms.

SECONDARY OUTCOMES:
Pain Level (Numerical Rating Scale) | 5 weeks
  Pain intensity will be self-assessed by adolescents using a 0-10 scale, where 0 represents no pain and 10 represents the worst possible pain. The change in pain levels will be tracked over the study.
Quality of Life (SF-36 Score) | 5 weeks
  uality of life will be assessed using the SF-36 Health Survey, which evaluates physical and mental health across eight domains. Higher scores indicate better health status.
Medication Consumption | 5 weeks
  This measure tracks changes in the quantity and dosage of medications used by participants for pain, somatic symptoms, or related conditions.
Anxiety and Depression (HAD Score) | 5 weeks
  Anxiety and depression levels will be assessed using the Hospital Anxiety and Depression (HAD) Scale, where higher scores reflect more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The Mondor Clinical Research Unit (URC Mondor), Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION